CLINICAL TRIAL: NCT02107196
Title: A 12-Week Double-blind, Randomised, Placebo-controlled, Parallel Group Phase III Study, Followed by a 4-Week Randomised Withdrawal Period to Evaluate the Efficacy and Safety of Oral Ibodutant 10 mg Once Daily in Female Patients With Irritable Bowel Syndrome With Diarrhea
Brief Title: 12-Week Efficacy and Safety Study of Ibodutant in Women With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Acronym: IRIS-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAK-06; 2013-000894-56 (EudraCT Number)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Results first posted 2016-09-27 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-11

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: Irritable Bowel Syndrome; Colon, irritable; Bowel disease; Diarrhea
MeSH Terms: conditions — Irritable Bowel Syndrome; Intestinal Diseases; Diarrhea | interventions — ibodutant; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibodutant 10 mg (Experimental): Oral tablet to be given once daily for 12 weeks of treatment. Patients randomised to the ibodutant 10 mg arm will be re-randomised at week 13 in a 1:1 ratio to either ibodutant 10 mg or placebo for additional 4 weeks of treatment.
  Interventions: Drug: Ibodutant 10 mg
- Placebo (Placebo Comparator): Oral tablet to be given once daily for 12 weeks of treatment. Patients randomised to the placebo arm will be mock-re-randomised (switch in blinded conditions) to ibodutant at week 13 for additional 4 weeks of treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibodutant 10 mg — Oral tablet, to be given once daily.
  Other Names: Code: MEN 15596
  Arms: Ibodutant 10 mg
Drug: Placebo — Oral tablet, (identical in appearance and weight to ibodutant tablets), to be given once daily.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Irritable Bowel Syndrome with diarrhoea (IBS-D) is a functional gastrointestinal disorder characterised by chronic or recurrent abdominal pain or discomfort and diarrhoea. This trial aims at the evaluation of the efficacy and safety of oral ibodutant 10 mg once daily as compared to placebo in women with IBS-D over a 12-week treatment period.

DETAILED DESCRIPTION:
The study evaluates the efficacy and safety of ibodutant 10 mg, given once daily for 12 weeks in comparison with placebo in female IBS-D patients. Randomisation to ibodutant and placebo will be 1:1. Efficacy is evaluated in terms of weekly response for abdominal pain intensity and stool consistency over 12 weeks of treatment in at least 50% of the weeks of treatment.

The clinical phase of the study comprises up to 2 weeks of screening for patient's eligibility, a 2-week run-in period (treatment-free) for IBS severity assessment, a 12-week double-blind treatment period, a 4-week randomised withdrawal (RW) period and a 2-week safety follow-up, resulting in a maximum 22-week overall duration of the study for each patient.

Patients report their IBS-related symptoms daily in a telephone-based electronic diary from run-in until end of treatment.

ELIGIBILITY:
Inclusion Criteria:

At screening:

* Female patients aged 18 years or older.
* Clinical diagnosis of IBS-D according to the following symptoms-based criteria as per Rome III modular questionnaire criteria:

  1. Recurrent abdominal pain or discomfort for at least 3 days per month in the last 3 months associated with at least 2 of the following characteristics: a) improvement with defecation; b) onset associated with a change in the frequency of stool; c) onset associated with a change in form (appearance) of stool.
  2. Symptom-onset at least 6 months prior to diagnosis.
  3. Loose or watery stools at least 25% of the time in the last 3 months AND hard or lumpy stools less than 25% of the time in the last 3 months.
  4. Additional criterion: more than 3 bowel movements per day at least 25% of the time in the last 3 months.
* For patients older than 50 years OR patients with a positive family history of colorectal cancer: normal results from colonoscopy/flexible sigmoidoscopy performed within the last 5 years.
* For patients aged 65 years or older: absence of ischaemic colitis, microscopy colitis or any other organic gastrointestinal disease as evidenced by the results of a colonoscopy/flexible sigmoidoscopy with biopsy performed within 6 months.
* For women of childbearing potential: Use of a highly effective contraceptive method with a failure rate <1% per year throughout the entire study period.
* Physical examination without clinically relevant abnormalities during screening.
* No clinically relevant abnormalities in 12-Lead ECG or in laboratory findings.
* Mentally competent, able to give written informed consent, and compliant to undergo all visits and procedures.
* Unrestricted access to a touch-tone telephone.
* Willingness to refrain from using loperamide within 3 days prior to run-in visit and during the run-in period.

Additional criteria at randomisation:

* During both weeks of the run-in period:

  1. A weekly average of worst abdominal pain in the past 24 hours with a score of ≥3.0 on a 0 to 10 point scale.
  2. At least one bowel movement on each day.
  3. A weekly average of at least 3 bowel movements per day.
  4. At least one stool with a consistency of Type 6 or Type 7 according to the Bristol Stool Scale (BSS) on at least 2 days per week.
  5. Less than 2 bowel movements with a consistency of Type 1 or Type 2 according to the BSS per week.
* Adequate compliance with the e-diary recording procedure defined as at least 11 of 14 days (≥75%) of the nominal daily data entry.

Exclusion Criteria:

* Male gender.
* Diagnosis of IBS with a subtype of constipation, mixed IBS, or un-subtyped IBS.
* Colonic or major abdominal surgery, any other major abdominal surgery or elective major surgery planned or expected during the study.
* History of organic GI abnormalities, inflammatory bowel diseases, complicated diverticulosis, ischaemic colitis, microscopic colitis.
* History of pancreatitis, active biliary duct disease, cholecystitis or symptomatic gallbladder stone disease in the previous 6 months.
* History of gluten enteropathy or lactose intolerance.
* Current or previous diagnosis of neoplasia.
* History of endometriosis.
* History of positive tests for ova or parasites, or clostridium difficile toxin or occult blood in the stool in the previous 6 months.
* History of human immunodeficiency virus infection.
* History of major cardiovascular events in the previous 6 months.
* Uncontrolled hypertension, insulin-dependent diabetes mellitus or abnormal thyroid function.
* Major psychiatric or neurological disorders or unstable medical condition which may compromise the efficacy and safety assessments.
* Evidence of clinically significant hepatic disease, severe renal insufficiency or anemia.
* Relevant changes in dietary habits, lifestyle, or exercise regimen in the previous 2 months.
* Use of prohibited concurrent medication within the previous month such as antibiotics, antimuscarinic drugs, drugs enhancing GI motility and analgesics.
* Pregnancy or breastfeeding.
* Inability to understand or collaborate throughout the study.
* Participation in other clinical studies in the previous 4 weeks or concurrent enrollment in a clinical study.
* Any condition that would compromise the well-being of the patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan F Tack, Professor, Study Chair — Department of Gastroenterology, University Hospital Gasthuisberg, Katholieke Universiteit Leuven, Leuven, Belgium; Lin Chang, Professor, Study Chair — Digestive Health and Nutrition Clinic. University of California, Los Angeles, CA, USA
Locations (110):
- United States (59):
  - Huntsville, Alabama
  - Sherwood, Arizona
  - Little Rock, Arkansas
  - Artesia, California
  - Chula Vista, California
  - Encino, California
  - Mission Hills, California
  - Sacramento, California
  - San Diego, California
  - Upland, California
  - Littleton, Colorado
  - Bristol, Connecticut
  - Boynton Beach, Florida
  - Brandon, Florida
  - Brooksville, Florida
  - Coral Gables, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Jupiter, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - Addison, Illinois
  - Chicago, Illinois
  - Augusta, Kansas
  - Newton, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Madisonville, Kentucky
  - Owensboro, Kentucky
  - Crowley, Louisiana
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Chesterfield, Michigan
  - Saginaw, Michigan
  - Troy, Michigan
  - Las Vegas, Nevada
  - Hartsdale, New York
  - Fayetteville, North Carolina
  - Greensboro, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Reading, Pennsylvania
  - Greer, South Carolina
  - Simpsonville, South Carolina
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Smyrna, Tennessee
  - Beaumont, Texas
  - Houston, Texas
  - Hurst, Texas
  - San Antonio, Texas
  - Ste. Channelview, Texas
  - West Jordan, Utah
  - Morgantown, West Virginia
- Bulgaria (5):
  - Haskovo
  - Plovdiv
  - Rousse
  - Sofia
  - Veliko Tarnovo
- Czechia (4):
  - Karlovy Vary
  - Prague
  - Ústí nad Labem
  - Ústí nad Orlicí
- France (5):
  - Bordeaux
  - Nantes
  - Nice
  - Rouen
  - Bobigny, Île-de-France Region
- Germany (4):
  - Stuttgart, Baden-Wurttemberg
  - Berlin
  - Essen
  - Hamburg
- Italy (5):
  - Bari
  - Bologna
  - Florence
  - Pavia
  - Rome
- Poland (5):
  - Bydgoszcz
  - Częstochowa
  - Krakow
  - Lublin
  - Wroclaw
- Romania (5):
  - Târgu Mureş, Jud. Mures
  - Târgu Mureş, Mureș County
  - Timișoara, Timiș County
  - Brasov
  - Bucharest
- Russia (5):
  - Kaluga
  - Moscow
  - Saint Petersburg
  - Smolensk
  - Yaroslavl
- Spain (6):
  - Badalona, Barcelona
  - Mataró, Barcelona
  - Sabadell, Barcelona
  - Barcelona
  - Madrid
  - Seville
- United Kingdom (7):
  - Penzance, Cornwall
  - Chesterfield, Derbyshire
  - Inverness, Scotland
  - Doncaster, South Yorkshire
  - Leicestershire
  - Manchester
  - Plymouth, Devon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was screened on 27th February 2014 and the first patient randomized on 21st March 2014. The last patient completed the study on 22nd June 2015. The study was conducted at 158 clinical sites in 11 countries (Bulgaria, Czech Republic, France, Germany, Italy, Poland, Romania, Russia, Spain, the USA and the United Kingdom).
Pre-assignment Details: A total of 1237 patients entered a 2-week Screening period, 1034 entered the qualifying 2-week Run-in period and 535 of them were randomised. After completion of the double-blind 12-week treatment, 453 patients entered into the Randomised Withdrawal (RW) period.
Groups:
- Ibodutant 10 mg: Oral tablet to be given once daily for 12 weeks of treatment. Patients randomized to the ibodutant 10 mg arm will be re-randomized at week 13 in a 1:1 ratio to either ibodutant 10 mg or placebo for additional 4 weeks of treatment.
  Ibodutant 10 mg: Oral tablet, to be given once daily.
- Placebo: Oral tablet to be given once daily for 12 weeks of treatment. Patients randomized to the placebo arm will be mock-re-randomized (switch in blinded conditions) to ibodutant at week 13 for additional 4 weeks of treatment.
  Placebo: Oral tablet, (identical in appearance and weight to ibodutant tablets), to be given once daily.
Period: 12-week Treatment Period
Arm/Group | Ibodutant 10 mg | Placebo
Started | 271 (Safety population, all enrolled patients who received at least one dose of study drug) | 264 (Safety population, all enrolled patients who received at least one dose of study drug)
Intention To Treat (ITT) | 271 (All randomised patients who took at least one dose of study drug during 12-week treatment period) | 264 (All randomised patients who took at least one dose of study drug during 12-week treatment period)
Modified ITT | 221 (All ITT patients, excluding patients of two sites (serious breach of GCP, disqualified Investigator)) | 216 (All ITT patients, excluding patients of two sites (serious breach of GCP, disqualified Investigator))
Completed | 227 | 225
Not Completed | 44 | 39
Not completed — Adverse Event | 6 | 3
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 3 | 6
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 15 | 12
Not completed — Protocol Violation | 7 | 8
Not completed — Reason Missing | 11 | 8
Period: 4-week Randomized Withdrawal (RW) Period
Arm/Group | Ibodutant 10 mg | Placebo
Started | 338 (all re-randomized patients at Visit 6 [Day85]) | 114 (all re-randomized patients at Visit 6 [Day85])
RW Population | 338 (All re-randomized ITT patients,who received at least 1 dose of ibodutant during RW period) | 114 (All re-randomized ITT patients,who received at least 1 dose of placebo during RW period)
Modified RW Population | 272 (all RW patients, excluding patients of two sites (serious breach of GCP, disqualified Investigator)) | 90 (all RW patients, excluding patients of two sites (serious breach of GCP, disqualified Investigator))
Completed | 315 | 109
Not Completed | 23 | 5
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Reason Missing | 18 | 5

BASELINE CHARACTERISTICS:
Population: Baseline analysis was performed on the ITT population (n=535). The ITT population includes all randomised patients who took at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibodutant 10 mg | Placebo | Total
Number analyzed (Participants) | 271 | 264 | 535
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (12.81) | 43.8 (12.47) | 43.1 (12.65)
Gender [Count of Participants; unit: Participants]
  Female | 271 | 264 | 535
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 149 | 136 | 285
  Not Hispanic or Latino | 122 | 128 | 250
Region of Enrollment [Number; unit: participants]
  North America | 202 | 198 | 400
  Europe | 69 | 66 | 135
Abdominal Pain Severity Score [Number; unit: participants] — Worst abdominal pain on a 0 to 10 scale, where 0 corresponds to no pain and 10 corresponds to worst possible pain.
  participants
    <5 | 46 | 37 | 83
    >=5 to <8 | 176 | 187 | 363
    >=8 | 49 | 40 | 89
IBS-SSS Score [Number; unit: participants] — IBS-SSS score calculated from the questionnaire evaluating primarily the intensity of IBS symptoms during a 10-day period:abdominal pain, distension, stool frequency and consistency, and interference with life in general.The IBS-SSS calculates the sum of these 5 items each scored on a visual analog scale from 0 to 100.All four domains contribute equally to the total score, yielding a range of 0 to 500 to categorize patients into three severity groups:mild (below 175), moderate (175-300), and severe (above 300).
  participants
    Mild IBS (<175) | 2 | 6 | 8
    Moderate IBS (175 to <300) | 35 | 44 | 79
    Severe IBS (>=300) | 233 | 212 | 445
    Missing | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Weekly Response for Abdominal Pain Intensity AND Stool Consistency Over 12 Weeks of Treatment in at Least 50% of the Weeks of Treatment (6 Out of 12 Weeks).
Description: The patient will be considered a weekly responder if she meets both of the following criteria in the same week:
  * Abdominal pain response: decrease in weekly average of worst abdominal pain score in the past 24 hours of at least 30% compared with baseline;
  * Stool consistency response: decrease of at least 50% in the number of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline. The patients reported Bristol Stoll Chart score based on a 1 to 7 scale where 1 corresponds to hard stool and 7 corresponds to watery diarrhoea.
Time Frame: 12 weeks
Population: The primary efficacy analysis was performed on the modified ITT population (n=437): all patients included in the ITT population excluding patients from one site, where a potential serious breach of GCP was reported, and from another site, where disqualification proceedings against the Investigator were confirmed by the FDA.
Measure: Number; unit: Percentage of Responders
Arm/Group | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 221 | 216
Percentage of Responders | 35.7 | 34.7

2. Secondary Outcome: Weekly Response for Abdominal Pain Intensity Over 12 Weeks of Treatment in at Least 50% of the Weeks of Treatment (6 Out of 12 Weeks).
Description: The patient will be considered a weekly abdominal pain responder if she meets the following criterion:
  * Decrease in weekly average of worst abdominal pain score in the past 24 hours of at least 30% compared with baseline.
Time Frame: 12 weeks
Population: The secondary efficacy analysis was performed on the modified ITT population (n=437): all patients included in the ITT population excluding patients from one site, where a potential serious breach of GCP was reported, and from another site, where disqualification proceedings against the Investigator were confirmed by the FDA.
Measure: Number; unit: percentage of responders
Arm/Group | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 221 | 216
percentage of responders | 48.0 | 47.7

3. Secondary Outcome: Weekly Response for Stool Consistency Over 12 Weeks of Treatment in at Least 50% of the Weeks of Treatment (6 Out of 12 Weeks).
Description: The patient will be considered a weekly stool consistency responder if she meets the following criterion:
  * Decrease of at least 50% in the number of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline. The patients reported Bristol Stool Chart score based on a 1 to 7 scale where 1 corresponds to hard stool and 7 corresponds to watery diarrhoea.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of responders
Arm/Group | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 221 | 216
percentage of responders | 44.8 | 43.1

4. Secondary Outcome: Weekly Response for Relief of Overall IBS Signs and Symptoms Over 12 Weeks of Treatment in at Least 50% of the Weeks of Treatment (6 Out of 12 Weeks).
Description: The patient will be considered a weekly responder if she has an IBS degree-of-relief equal to "completely relieved/improved" or "considerably relieved/improved".
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of responders
Arm/Group | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 221 | 216
percentage of responders | 21.3 | 19.0

5. Secondary Outcome: Evaluation of Rebound Effects
Description: Comparison between average abdominal pain intensity (worst abdominal pain on a 0 to 10 NRS scale, where 0 corresponds to no pain and 10 corresponds to worst possible pain) and average stool consistency score (the patients reported Bristol Stool Chart score based on a 1 to 7 NRS scale where 1 corresponds to hard stool and 7 corresponds to watery diarrhoea) during the 4-week RW presented as change to baseline.
  The analysis only included the patients randomised to ibodutant in the 12-week treatment period and re-randomised to placebo for the 4-week RW period. Baseline was considered as the average abdominal pain intensity/stool consistency in the 2-week Run-in period.
Time Frame: 4 weeks
Population: modified RW population: only patients randomised to ibodutant in the 12-week treatment period and re-randomized to placebo for the 4-week RW period (excluding patients from one site, where a potential serious breach of GCP was reported, and another site, where disqualification proceedings against the Investigator were confirmed by FDA).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibodutant 10 mg
Number analyzed (Participants) | 89
units on a scale
  Baseline-Abdominal Pain Score (NRS, 0-10 points) | 6.53 (1.60)
  4-week RW-Abdominal Pain Score (NRS, 0-10 points) | -3.11 (2.21)
  Baseline-Bristol Stool Scale (NRS, 1 - 7 points) | 6.05 (0.52)
  4-week RW-Bristol Stool Scale (NRS, 1 - 7 points) | -1.38 (1.37)

ADVERSE EVENTS:
Time Frame: 12-week double blind treatment period
Arm/Group | Ibodutant 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/271 | 2/264
Other Adverse Events (participants affected / at risk) | 35/271 | 33/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibodutant 10 mg (N=271) | Placebo (N=264)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Circulatory Collaps (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibodutant 10 mg (N=271) | Placebo (N=264)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 7 (7) | 6 (6)
Urinary tract infections (Infections and infestations) | 8 (8) | 7 (8)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
muscle spasm (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting the results of this study for publication or presentation, the Investigator will allow the sponsor at least 30 days time to review and comment upon the publication manuscript. It is agreed, that the results of the study will not be submitted for presentation, abstract, poster exhibition, or publication by the investigator until Menarini Ricerche S.p.A. has reviewed/commented and agreed to any publication.